CLINICAL TRIAL: NCT02971930
Title: Exit Interviews to Assess Impact of Infusion Frequency in Hemophilia A
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19144
Record Dates: First submitted 2016-10-27; First posted 2016-11-23 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prophylaxis treatment of BAY94-9027_1: 2 infusions per week during the extension study
  Interventions: Biological: BAY94-9027
- Prophylaxis treatment of BAY94-9027_2: infusion every 5 days during the extension study
  Interventions: Biological: BAY94-9027
- Prophylaxis treatment of BAY94-9027_3: every 7 days during the extension study
  Interventions: Biological: BAY94-9027

INTERVENTIONS:
Biological: BAY94-9027 — Intravenous infusion of BAY94-9027

SUMMARY:
This study is to generate qualitative data to evaluate the impact of frequency of FVIII infusions on patients' satisfaction with treatment and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient is enrolled in the BAY94-9027 extension studies or is within 3 months of having completed participation in the BAY94-9027 extension studies;
* Patient allocated to Arm 2, Arm 3 or Arm 4 of BAY94-9027 extension studies.

  * Arm 2 Prophylaxis treatment of BAY94-9027; 2 infusions per week during the extension study
  * Arm 3 Prophylaxis treatment of BAY94-9027; infusion every 5 days during the extension study
  * Arm 4 Prophylaxis treatment of BAY94-9027; every 7 days during the extension study
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Patient must be willing and able to participate in a telephone interview lasting up to 30 minutes;
* Patient must have sufficient cognitive and linguistic capacities to allow them to actively participate in an interview lasting 30 minutes.

Exclusion Criteria:

* Patient is part of Arm 1: On-demand treatment of BAY94-9027 at individual dose and number of infusions based upon location and severity of bleeds;
* Patient is unlikely to comply with the study protocol (e.g. uncooperative attitude) or unlikely to complete the study for any reason in the opinion of the recruiter;
* Patient has great difficulty hearing or reading;
* Patient has any significant comorbid condition (including uncontrolled psychiatric conditions) that might limit or interfere with their ability to talk about their Hemophilia A and participate in the study;
* Patient has severe neurological or cognitive deficits that might affect their ability to participate in an interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients aged 18+ years who are participating in the BAY94-9027 extension studies or who are within 3 months of exiting the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Qualitative interviews (with patients) to determine patients' satisfaction | up to 4 months
  To conduct qualitative interviews with patients with Hemophilia A who have participated in the BAY94-9027 extension studies to evaluate patient experiences of and perspectives regarding their current treatment and the extent to which the frequency of FVIII infusions (compared to previous treatments) influences satisfaction
Qualitative interviews (with patients) to determine patients' quality of life | up to 4 months
  To conduct qualitative interviews with patients with Hemophilia A who have participated in the BAY94-9027 extension studies to evaluate patient experiences of and perspectives regarding their current treatment and the extent to which the frequency of FVIII infusions (compared to previous treatments) influences quality of life;
Qualitative interviews (with treating physicians) to determine patients' satisfaction | up to 4 months
  To conduct qualitative interview with clinicians who treat patients with Hemophilia A who have participated in the BAY94-9027 extension studies to evaluate the clinician perspective of patient experiences of and perspectives regarding their current treatment and the extent to which the frequency of FVIII infusions (compared to previous treatments) influences their patients' satisfaction
Qualitative interviews (with treating physicians) to determine patients' quality of life | up to 4 months
  To conduct qualitative interview with clinicians who treat patients with Hemophilia A who have participated in the BAY94-9027 extension studies to evaluate the clinician perspective of patient experiences of and perspectives regarding their current treatment and the extent to which the frequency of FVIII infusions (compared to previous treatments) influences their patients' quality of life;

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland, Cleveland, Ohio, United States